CLINICAL TRIAL: NCT07391995
Title: Evaluation of a New Diagnostic Tool (MinION) for Identifying Microorganisms in the Foot Wounds of Patients Living With Diabetic Foot Osteomyelitis (DFOM)
Brief Title: New Diagnostic Tool (MinION) for Identifying Microorganisms in Foot Wounds of Patients Living With Diabetic Foot Osteomyelitis
Acronym: MINI-OS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2025-1/MM-01
Record Dates: First submitted 2026-01-28; First posted 2026-02-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus; Diabetes Complications; Diabetic Peripheral Neuropathy
Keywords: Foot Ulcer, Diabetic; Infection
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Complications; Diabetic Foot; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 147 bone biopsies from 43 diabetic patients collected in the orthopaedic surgery operating theatre
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetic foot wound infections are predominantly polymicrobial. However, 'conventional' microbiological culture does not identify all the bacteria potentially involved in these infections and requires time, which can have a negative impact by delaying treatment and/or the prescription of appropriate antibiotic therapy.

Real-time metagenomics analysis using Oxford Nanopore Technologies' MinION technology has demonstrated sufficient power to identify virtually all microbial genomes in a given sample, providing additional information on their antibiotic resistance profile and in silico prediction of genes encoding virulence factors within than 4 hours. Based on these rapid results, a management protocol could be defined specifically for each patient with a view to personalised medicine.

The aim is to study the diversity of bacterial and fungal species identified using the MinION method and compare this diversity with the results obtained using conventional methods (routine culture) from bone biopsies taken from DFOM patients.

DETAILED DESCRIPTION:
Diabetes mellitus is one of the most common diseases in the world. Among its complications, 34% of patients living with diabetes will develop foot ulcers during their lifetime. Once this lesion has developed due to triopathy (arteriopathy, neuropathy, immunopathy), over 50% of these wounds will become infected, leading to serious consequences: bone damage (60 to 80% of cases), amputation (20% of infected wounds), mortality (68% at 5 years) and morbidity. The additional costs associated with this condition exceed $850 billion worldwide, with $1 million spent every 30 seconds due to complications from these wounds in the US. Diabetic foot ulcers (DFUs) are therefore a major public health problem.

For infectious disease specialists, one of the main difficulties in treating infections in these wounds is distinguishing between bacterial colonization - a physiological process, and infection - a pathological process. Studies of the microbiota of foot wounds in diabetic patients show the polymicrobial nature of these lesions, which contain commensal bacteria from the skin microbiota, opportunistic pathogenic bacteria and bacteria from the environment. Among Gram-positive cocci, Staphylococcus aureus is the species most often identified in diabetic foot osteomyelitis (DFO) (23.4%), followed by Pseudomonas spp. (11.1%), Escherichia coli (11.5%), Proteus spp. (8.3%), Klebsiella spp. (6.9%), and Enterococcus spp. (5.4%). Coagulase-negative staphylococci, although involved in less than 4% of infections, often remain difficult to identify by mass spectrometry at species level, even though some of them are known for their pathogenicity. The other major difficulty is the time it takes to obtain results when osteomyelitis is suspected. In such situations, obtaining a bone sample is the standard method and the best way to identify the pathogen(s) responsible and their sensitivity to antibiotics. Bone biopsy can be performed intraoperatively or percutaneously, as recommended by the International Working Group of the Diabetic Foot (IWGDF) in 2023. In addition, to avoid false-negative cultures, experts suggest delaying bone biopsy in patients already on antibiotics, ideally for at least two weeks. In the microbiology laboratory, the standard diagnosis based on conventional microbiological culture can take up to two weeks to identify the causative bacteria and perform antibiotic susceptibility testing on the responsible pathogen(s), bringing the total time to establish a diagnosis to 4 weeks.To reduce this delay, certain culture-free molecular microbiology techniques, in particular metagenomic next-generation sequencing (mNGS), have shown that the microbiota of most wound infections is more diverse and abundant than that revealed by conventional culture methods. However, very few metagenomic data on bone biopsies from DFOMs are available. As molecular biology tools were unable to distinguish between live and dead bacterial cells and cannot identify the bacterial genera contributing to the clinical status of the infection, their use in daily practice is not recommended by the IWGDF and SPILF (Société de Pathologie Infectieuse de Langue Française), as their results could lead to the unnecessary use of broad-spectrum antibiotics. Recent studies based on metagenomic analysis of bone biopsies, soft tissue biopsies and swabs from foot wounds in diabetic patients have identified microbial diversity as a marker of infection. The number of bacteria involved in confirmed cases of infection is estimated at over 70, a figure difficult to achieve with conventional routine methods. The use of PCR based on amplification of the gene coding for 16S rRNA is considered unsuitable due to the frequent polymicrobial nature of DFOM samples. Multiplex PCR methods are not exhaustive in identifying all pathogens. Finally, conventional culture methods are often time-consuming, and species identification using laboratory methods such as MALDI-TOF mass spectrometry is often a source of confusion or failure. Recently, a new rapid sequencing tool has been developed: the MinION. It is small and fast and can sequence a bacterial or viral genome from single-microbe samples in less than four hours, or determine a panel of microorganisms present in a more complex sample. This tool is particularly useful for cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 147 bone biopsies from 43 diabetic patients collected in the orthopedic surgery operating room
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of bacterial and fungal species found in a conventional bone biopsy | 12 months
  Number of species found by each method (presence/absence and species identification): bacterial and fungal species detected in bone biopsies by the two methods (conventional culture vs MinION
Number of bacterial and fungal species found with the MiniON device | 12 months
  Number of species found by each method (presence/absence and species identification): bacterial and fungal species detected in bone biopsies by the two methods (conventional culture vs MinION

SECONDARY OUTCOMES:
Description of the bone microbiota of diabetic foot osteomyelitis using the MinION method | 12 months
  Typology of microbial species found using the MinION method. The MinION™ Mk1D is the next generation of portable nanopore sequencing devices. Improved thermal dissipation capabilities of the MinION Mk1D significantly enhances sequencing performance, enabling highly accurate real-time sequencing in an even wider range of environments than its predecessor, the MinION Mk1B.
Description of the bone microbiota of diabetic foot osteomyelitis using the conventional method (MALDI-TOF) | 12 months
  Typology of microbial species found using the MALDI-TOF method. The MALDI-TOF (Matrix Assisted Laser Desorption Ionization - Time of Flight) instrument is a mass spectrometer that combines a matrix-assisted laser ionization source (MALDI) with a time-of-flight analyzer (TOF). One of the important characteristics of mass spectrometry is peak sharpness, measured by the resolution of the mass spectrometer. Resolution is defined as the ratio of the peak mass m to the full width at half maximum Δm. The higher the resolution, the sharper the peaks. This makes it possible to visualize two molecules with similar masses. MALDI-TOF instruments can be equipped with a reflection (electrostatic mirror or "ion mirror") that deflects ions with an electric field, thereby doubling the length of the ion flight path and increasing the resolution of the instrument. A MALDI-TOF mass spectrometer can achieve resolutions of 5000 in linear mode (without reflection) and 20000 with reflecton.
New potentially pathogenic species in diabetic foot osteomyelitis in relation to wound progression. | 3 months
  Degree of wound healing at 3 months, 6 months and one year, depending on the presence or absence of different microbial species.
New potentially pathogenic species in diabetic foot osteomyelitis in relation to wound progression. | 6 months
  Degree of wound healing at 3 months, 6 months and one year, depending on the presence or absence of different microbial species.
New potentially pathogenic species in diabetic foot osteomyelitis in relation to wound progression. | 12 months
  Degree of wound healing at 3 months, 6 months and one year, depending on the presence or absence of different microbial species.
Antibiotic sensitivity profiles of microorganisms obtained in vitro (bacterial culture). | 12 months
  The number and % of strains resistant to antibiotics tested on pathogenic bacteria isolated in standard microbiological culture will be recorded.
Antibiotic sensitivity profiles of microorganisms obtained in silico (MinION technology). | 12 months
  Presence/absence of resistance genes to the antibiotic families tested on pathogenic bacteria isolated in standard microbiological culture
Cost of conventional in vitro culture and testing | 12 months
  Cost in Euros
Cost of using in silico MinION technology | 12 months
  Cost in Euros

OTHER OUTCOMES:
Gender of patients providing samples | Baseline
  Male/female/Non-binary
Age of patients providing samples | Baseline
  In years
Body mass index of patients providing samples | Baseline
  The formula is BMI = kg/m2; kg is a person's weight in kilograms and m2 is height in meters squared
Wound grade | Baseline
  Wagner Grade 1: Partial- or full-thickness ulcer (superficial ulcer) Wagner Grade 2: Deep ulcer extended to ligament, tendon, joint capsule, bone, or deep fascia without abscess or osteomyelitis (OM) Wagner Grade 3: Deep abscess, OM, or joint sepsis. Wagner Grade 4: Partial-foot gangrene.
Previous antibiotherapy | Baseline
  YES/NO
Evolution of the wound at 3 months | Month 3
  Healed/Worsening
Evolution of the wound at 6 months | Month 6
  Healed/Worsening
Evolution of the wound at 12 months | Month 12
  Healed/Worsening

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Dubois, Dr., Principal Investigator — Nîmes University Hospital
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France

REFERENCES:
- [Background] Lipsky BA, Senneville E, Abbas ZG, Aragon-Sanchez J, Diggle M, Embil JM, Kono S, Lavery LA, Malone M, van Asten SA, Urbancic-Rovan V, Peters EJG; International Working Group on the Diabetic Foot (IWGDF). Guidelines on the diagnosis and treatment of foot infection in persons with diabetes (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3280. doi: 10.1002/dmrr.3280. PMID 32176444
- [Background] Cascini S, Agabiti N, Davoli M, Uccioli L, Meloni M, Giurato L, Marino C, Bargagli AM. Survival and factors predicting mortality after major and minor lower-extremity amputations among patients with diabetes: a population-based study using health information systems. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001355. doi: 10.1136/bmjdrc-2020-001355. PMID 32690575
- [Background] Armstrong DG, Kanda VA, Lavery LA, Marston W, Mills JL Sr, Boulton AJ. Mind the gap: disparity between research funding and costs of care for diabetic foot ulcers. Diabetes Care. 2013 Jul;36(7):1815-7. doi: 10.2337/dc12-2285. No abstract available. PMID 23801792
- [Background] Radzieta M, Sadeghpour-Heravi F, Peters TJ, Hu H, Vickery K, Jeffries T, Dickson HG, Schwarzer S, Jensen SO, Malone M. A multiomics approach to identify host-microbe alterations associated with infection severity in diabetic foot infections: a pilot study. NPJ Biofilms Microbiomes. 2021 Mar 22;7(1):29. doi: 10.1038/s41522-021-00202-x. PMID 33753735
- [Background] Jneid J, Cassir N, Schuldiner S, Jourdan N, Sotto A, Lavigne JP, La Scola B. Exploring the Microbiota of Diabetic Foot Infections With Culturomics. Front Cell Infect Microbiol. 2018 Aug 14;8:282. doi: 10.3389/fcimb.2018.00282. eCollection 2018. PMID 30155447
- [Background] Macdonald KE, Boeckh S, Stacey HJ, Jones JD. The microbiology of diabetic foot infections: a meta-analysis. BMC Infect Dis. 2021 Aug 9;21(1):770. doi: 10.1186/s12879-021-06516-7. PMID 34372789
- [Background] Manas AB, Taori S, Ahluwalia R, Slim H, Manu C, Rashid H, Kavarthapu V, Edmonds M, Vas PRJ. Admission Time Deep Swab Specimens Compared With Surgical Bone Sampling in Hospitalized Individuals With Diabetic Foot Osteomyelitis and Soft Tissue Infection. Int J Low Extrem Wounds. 2021 Dec;20(4):300-308. doi: 10.1177/1534734620916386. Epub 2020 May 5. PMID 32370639
- [Background] Macauley M, Adams G, Mackenny P, Kubelka I, Scott E, Buckworth R, Biddiscombe C, Aitkins C, Lake H, Matthews V, Ashraff S, Ashwell S. Microbiological evaluation of resection margins of the infected diabetic foot ulcer. Diabet Med. 2021 Apr;38(4):e14440. doi: 10.1111/dme.14440. Epub 2020 Nov 11. PMID 33113230
- [Background] Senneville E, Albalawi Z, van Asten SA, Abbas ZG, Allison G, Aragon-Sanchez J, Embil JM, Lavery LA, Alhasan M, Oz O, Uckay I, Urbancic-Rovan V, Xu ZR, Peters EJG. IWGDF/IDSA guidelines on the diagnosis and treatment of diabetes-related foot infections (IWGDF/IDSA 2023). Diabetes Metab Res Rev. 2024 Mar;40(3):e3687. doi: 10.1002/dmrr.3687. Epub 2023 Oct 1. PMID 37779323
- [Background] Chen Y, Shi Y, Zhu W, You J, Yang J, Xie Y, Zhao H, Li H, Fan S, Li L, Liu C. Combining CRISPR-Cas12a-Based Technology and Metagenomics Next Generation Sequencing: A New Paradigm for Rapid and Full-Scale Detection of Microbes in Infectious Diabetic Foot Samples. Front Microbiol. 2021 Oct 7;12:742040. doi: 10.3389/fmicb.2021.742040. eCollection 2021. PMID 34690988
- [Background] Malone M, Johani K, Jensen SO, Gosbell IB, Dickson HG, Hu H, Vickery K. Next Generation DNA Sequencing of Tissues from Infected Diabetic Foot Ulcers. EBioMedicine. 2017 Jul;21:142-149. doi: 10.1016/j.ebiom.2017.06.026. Epub 2017 Jun 27. PMID 28669650
- [Background] Morsli M, Salipante F, Magnan C, Dunyach-Remy C, Sotto A, Lavigne JP. Direct metagenomics investigation of non-surgical hard-to-heal wounds: a review. Ann Clin Microbiol Antimicrob. 2024 May 3;23(1):39. doi: 10.1186/s12941-024-00698-z. PMID 38702796
- [Background] Eshaghi A, Bommersbach C, Zittermann S, Burnham CA, Patel R, Schuetz AN, Patel SN, Kus JV. Phenotypic and Genomic Profiling of Staphylococcus argenteus in Canada and the United States and Recommendations for Clinical Result Reporting. J Clin Microbiol. 2021 May 19;59(6):e02470-20. doi: 10.1128/JCM.02470-20. Print 2021 May 19. PMID 33731414
- [Background] Morsli M, Bechah Y, Coulibaly O, Toro A, Fournier PE, Houhamdi L, Drancourt M. Direct diagnosis of Pasteurella multocida meningitis using next-generation sequencing. Lancet Microbe. 2022 Jan;3(1):e6. doi: 10.1016/S2666-5247(21)00277-9. Epub 2021 Nov 11. No abstract available. PMID 35544115
- [Background] Morsli M, Kerharo Q, Amrane S, Parola P, Fournier PE, Drancourt M. Real-time whole genome sequencing direct diagnosis of Streptococcus pneumoniae meningitis: A case report. J Infect. 2021 Dec;83(6):709-737. doi: 10.1016/j.jinf.2021.10.002. Epub 2021 Oct 8. No abstract available. PMID 34627841
- [Background] Morsli M, Boudet A, Kerharo Q, Stephan R, Salipante F, Dunyach-Remy C, Houhamdi L, Fournier PE, Lavigne JP, Drancourt M. Real-time metagenomics-based diagnosis of community-acquired meningitis: A prospective series, southern France. EBioMedicine. 2022 Oct;84:104247. doi: 10.1016/j.ebiom.2022.104247. Epub 2022 Sep 7. PMID 36087524
- See also: Link to IDF Diabetes Atlas — http://www.diabetesatlas.org/